CLINICAL TRIAL: NCT01165177
Title: Efficacy, Safety, and Immunogenicity Study of GSK Biologicals' Herpes Zoster Vaccine GSK1437173A in Adults Aged 50 Years or Older
Brief Title: Study to Evaluate Efficacy, Safety and Immunogenicity of GSK Biologicals' Herpes Zoster (HZ) Vaccine GSK1437173A in Adults Aged 50 Years and Older
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 110390; 2008-000367-42 (EudraCT Number)
Record Dates: First submitted 2010-07-15; First posted 2010-07-19 (Estimated); Results first posted 2017-05-01 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-01

CONDITIONS: Herpes Zoster
Keywords: subjects 50 years and older; vaccine; immunogenicity; efficacy; Herpes Zoster; safety
MeSH Terms: conditions — Herpes Zoster

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- GSK1437173A group (Experimental): Subjects will receive Herpes Zoster Vaccine GSK1437173A according to a 0, 2-month schedule
  Interventions: Biological: Herpes Zoster Vaccine GSK1437173A
- Placebo group (Placebo Comparator): Subjects will receive NaCl solution placebo according to a 0, 2-month schedule
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Herpes Zoster Vaccine GSK1437173A — Intramuscular injection
  Arms: GSK1437173A group
Biological: Placebo — Intramuscular injection
  Arms: Placebo group

SUMMARY:
The purpose of this observer-blind study is to evaluate the efficacy, safety and immunogenicity of GSK Biologicals' candidate Herpes Zoster (HZ) vaccine in adults aged ≥ 50 years.

Two studies [ZOSTER-006 (NCT01165177) and ZOSTER-022 (NCT01165229)] are being conducted concurrently to evaluate efficacy of GSK1437173A vaccine. A pooled analysis of data from both studies combined will be conducted contingent on each study achieving its objectives. The protocol posting of study ZOSTER-022 also deals with the outcome measures related to the pooled analysis.

DETAILED DESCRIPTION:
This protocol summary has been updated following Protocol Amendment 4 changes to study objectives and endpoints and the analyses of the objectives in 2 steps.

Step 1 will include analyses of the following objectives of ZOSTER-006 (NCT01165177): all HZ VE objectives and all reactogenicity/safety and immunogenicity objectives. At step 2, all objectives of study ZOSTER-006 (NCT01165177) will be analyzed. Objectives already analyzed at step 1 will be re-analyzed (confirmatory descriptive in case of inferential analysis at step 1 or descriptive analysis otherwise). At step 2, pooled analyses of studies ZOSTER-006 (NCT01165177) and ZOSTER-022 (NCT01165229) are planned; overall PHN VE in subjects ≥ 70 YOA, and other pre-specified endpoints will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes will comply with the requirements of the protocol;
* Written informed consent obtained from the subject;
* A male or female aged 50 years or older at the time of the first vaccination;
* Female subjects of non-childbearing potential may be enrolled in the study;

For this study population, non-childbearing potential is defined as current tubal ligation, hysterectomy, ovariectomy or post-menopause.

OR Female subjects of childbearing potential may be enrolled in the study, if the subject has practiced adequate contraception for 30 days prior to vaccination, and has a negative urine pregnancy test on the day of vaccination, and has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series;

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period;
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product;
* Any confirmed or suspected immunosuppressive or immunodeficient condition resulting from disease or immunosuppressive/cytotoxic therapy;
* History of HZ;
* Previous vaccination against varicella or HZ;
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine. Additionally, consider allergic reactions to other material or equipment related to study participation;
* Significant underlying illness that in the opinion of the investigator would be expected to prevent completion of the study;
* Receipt of immunoglobulins and/or any blood products within the 90 days preceding the first dose of study vaccine or planned administration during the study period;
* Administration or planned administration of any other immunizations within 30 days before the first or second study vaccination or scheduled within 30 days after study vaccination. However, licensed non-replicating vaccines may be administered up to 8 days prior to each dose and/or at least 14 days after any dose of study vaccine;
* Any other condition that, in the opinion of the investigator, might interfere with the evaluations required by the study;
* Acute disease and/or fever at the time of enrollment;
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Pregnant or lactating female;
* Female planning to become pregnant or planning to discontinue contraceptive precautions.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16165 (Actual)
Dates: Start 2010-08-02 (Actual); Primary Completion 2014-05-09 (Actual); Study Completion 2015-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (184):
- United States (39):
  - GSK Investigational Site, Mesa, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Spring Valley, California
  - GSK Investigational Site, Vista, California
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, DeLand, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Meridian, Idaho
  - GSK Investigational Site, Overland Park, Kansas
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Columbia, Maryland
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Edison, New Jersey
  - GSK Investigational Site, Somers Point, New Jersey
  - GSK Investigational Site, Cary, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Hickory, North Carolina
  - GSK Investigational Site, Salisbury, North Carolina
  - GSK Investigational Site, Wilmington, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Wadsworth, Ohio
  - GSK Investigational Site, Carnegie, Pennsylvania
  - GSK Investigational Site, Pleasant Hills, Pennsylvania
  - GSK Investigational Site, Uniontown, Pennsylvania
  - GSK Investigational Site, Greer, South Carolina
  - GSK Investigational Site, Mt. Pleasant, South Carolina
  - GSK Investigational Site, Bristol, Tennessee
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Murray, Utah
  - GSK Investigational Site, Arlington, Virginia
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Winchester, Virginia
  - GSK Investigational Site, Renton, Washington
- Australia (8):
  - GSK Investigational Site, Glebe, New South Wales
  - GSK Investigational Site, Maroubra, New South Wales
  - GSK Investigational Site, Umina, New South Wales
  - GSK Investigational Site, Westmead, New South Wales
  - GSK Investigational Site, Wollongong, New South Wales
  - GSK Investigational Site, Sherwood, Queensland
  - GSK Investigational Site, Geelong, Victoria
  - GSK Investigational Site, Ivanhoe, Victoria
- Brazil (5):
  - GSK Investigational Site, Belo Horizonte, Minas Gerais
  - GSK Investigational Site, Curitiba/Paraná, Paraná
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
  - GSK Investigational Site, Curitiba/PR
  - GSK Investigational Site, São Paulo
- Canada (13):
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Victoria, British Columbia
  - GSK Investigational Site, Bay Roberts, Newfoundland and Labrador
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Woodstock, Ontario
  - GSK Investigational Site, Gatineau, Quebec
  - GSK Investigational Site, Mirabel, Quebec
  - GSK Investigational Site, Pointe-Claire, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
  - GSK Investigational Site, Trois-Rivières, Quebec
- Czechia (3):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, České Budějovice
  - GSK Investigational Site, Hradec Králové
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- Finland (9):
  - GSK Investigational Site, Espoo
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Jarvenpaa
  - GSK Investigational Site, Kokkola
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Pori
  - GSK Investigational Site, Seinäjoki
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
- France (13):
  - GSK Investigational Site, Angers
  - GSK Investigational Site, Château-Gontier
  - GSK Investigational Site, Cherbourg
  - GSK Investigational Site, Clermont-Ferrand
  - GSK Investigational Site, Laval
  - GSK Investigational Site, Montrevault
  - GSK Investigational Site, Muret
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Rosiers-d'Égletons
  - GSK Investigational Site, Saint Cyr Sur Loir
  - GSK Investigational Site, Segré
  - GSK Investigational Site, Soulaines-sur-Aubance
  - GSK Investigational Site, Tours
- Germany (31):
  - GSK Investigational Site, Deggingen, Baden-Wurttemberg
  - GSK Investigational Site, Güglingen, Baden-Wurttemberg
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Tübingen, Baden-Wurttemberg
  - GSK Investigational Site, Wangen, Baden-Wurttemberg
  - GSK Investigational Site, Weinheim, Baden-Wurttemberg
  - GSK Investigational Site, Dachau, Bavaria
  - GSK Investigational Site, Künzing, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Rednitzhembach, Bavaria
  - GSK Investigational Site, Wallerfing, Bavaria
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Potsdam, Brandenburg
  - GSK Investigational Site, Flörsheim, Hesse
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Duelmen, Lower Saxony
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Goch, North Rhine-Westphalia
  - GSK Investigational Site, Witten, North Rhine-Westphalia
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Rhaunen, Rhineland-Palatinate
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Freiberg, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Pirna, Saxony
  - GSK Investigational Site, Köthen, Saxony-Anhalt
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Hong Kong (2):
  - GSK Investigational Site, Kwun Tong
  - GSK Investigational Site, Shatin
- Italy (11):
  - GSK Investigational Site, Chieti, Abruzzo
  - GSK Investigational Site, Pescara, Abruzzo
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Monza, Lombardy
  - GSK Investigational Site, Cuneo, Piedmont
  - GSK Investigational Site, Cagliari, Sardinia
  - GSK Investigational Site, Sassari, Sardinia
  - GSK Investigational Site, Catania, Sicily
  - GSK Investigational Site, Ragusa (RG), Sicily
- Japan (4):
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Tokyo
- Mexico (4):
  - GSK Investigational Site, Zapopan, Jalisco, Jalisco
  - GSK Investigational Site, Cuernavaca, Morelos
  - GSK Investigational Site, Durango
  - GSK Investigational Site, Monterrey
- South Korea (6):
  - GSK Investigational Site, Ansan
  - GSK Investigational Site, Bucheon-si
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Kangnam-gu, Seoul
  - GSK Investigational Site, Kangwon-do
  - GSK Investigational Site, Seoul
- Spain (10):
  - GSK Investigational Site, Alcover( Tarragona)
  - GSK Investigational Site, Balenyà (Barcelona)
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Centelles
  - GSK Investigational Site, La Roca Del Valles (Barcelona)
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Majadahonda
  - GSK Investigational Site, Peralada( Girona)
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Vic/ Barcelona
- Sweden (12):
  - GSK Investigational Site, Borås
  - GSK Investigational Site, Eskilstuna
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Jönköping
  - GSK Investigational Site, Karlskrona
  - GSK Investigational Site, Linköping
  - GSK Investigational Site, Malmo
  - GSK Investigational Site, Örebro
  - GSK Investigational Site, Skövde
  - GSK Investigational Site, Stockholm
  - GSK Investigational Site, Uppsala
  - GSK Investigational Site, Vällingby
- Taiwan (3):
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Taoyuan District
- United Kingdom (9):
  - GSK Investigational Site, Buckshaw Village, Chorley, Lancashire
  - GSK Investigational Site, Atherstone, Warwickshire
  - GSK Investigational Site, Bradford-on-Avon, Wiltshire
  - GSK Investigational Site, Bangor
  - GSK Investigational Site, Belfast
  - GSK Investigational Site, Broughshane
  - GSK Investigational Site, Ledbury
  - GSK Investigational Site, Newtonabbey
  - GSK Investigational Site, Waterloo, Liverpool

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Background] Cunningham AL, Lal H, Kovac M, Chlibek R, Hwang SJ, Diez-Domingo J, Godeaux O, Levin MJ, McElhaney JE, Puig-Barbera J, Vanden Abeele C, Vesikari T, Watanabe D, Zahaf T, Ahonen A, Athan E, Barba-Gomez JF, Campora L, de Looze F, Downey HJ, Ghesquiere W, Gorfinkel I, Korhonen T, Leung E, McNeil SA, Oostvogels L, Rombo L, Smetana J, Weckx L, Yeo W, Heineman TC; ZOE-70 Study Group. Efficacy of the Herpes Zoster Subunit Vaccine in Adults 70 Years of Age or Older. N Engl J Med. 2016 Sep 15;375(11):1019-32. doi: 10.1056/NEJMoa1603800. PMID 27626517
- [Background] Cunningham AL, Heineman TC, Lal H, Godeaux O, Chlibek R, Hwang SJ, McElhaney JE, Vesikari T, Andrews C, Choi WS, Esen M, Ikematsu H, Choma MK, Pauksens K, Ravault S, Salaun B, Schwarz TF, Smetana J, Abeele CV, Van den Steen P, Vastiau I, Weckx LY, Levin MJ; ZOE-50/70 Study Group. Immune Responses to a Recombinant Glycoprotein E Herpes Zoster Vaccine in Adults Aged 50 Years or Older. J Infect Dis. 2018 May 5;217(11):1750-1760. doi: 10.1093/infdis/jiy095. PMID 29529222
- [Background] Ikematsu H et al. (2018) Efficacy, safety and immunogenicity of new adjuvanted herpes zoster subunit vaccine for Japanese over 50 years old and over 70 years old. Kansenshogaku Zasshi. 92(2):103-114.
- [Background] Kovac M, Lal H, Cunningham AL, Levin MJ, Johnson RW, Campora L, Volpi A, Heineman TC; ZOE-50/70 Study Group. Complications of herpes zoster in immunocompetent older adults: Incidence in vaccine and placebo groups in two large phase 3 trials. Vaccine. 2018 Mar 14;36(12):1537-1541. doi: 10.1016/j.vaccine.2018.02.029. Epub 2018 Feb 17. PMID 29463421
- [Background] Lal H, Cunningham AL, Godeaux O, Chlibek R, Diez-Domingo J, Hwang SJ, Levin MJ, McElhaney JE, Poder A, Puig-Barbera J, Vesikari T, Watanabe D, Weckx L, Zahaf T, Heineman TC; ZOE-50 Study Group. Efficacy of an adjuvanted herpes zoster subunit vaccine in older adults. N Engl J Med. 2015 May 28;372(22):2087-96. doi: 10.1056/NEJMoa1501184. Epub 2015 Apr 28. PMID 25916341
- [Derived] Matthews S, Curran D, Sabater Cabrera E, Boutry C, Lecrenier N, Cunningham AL, Schmader K. An Analysis of How Herpes Zoster Pain Affects Health-related Quality of Life of Placebo Patients From 3 Randomized Phase III Studies. Clin J Pain. 2023 Aug 1;39(8):386-393. doi: 10.1097/AJP.0000000000001129. PMID 37166199
- [Derived] Kim JH, Johnson R, Kovac M, Cunningham AL, Amakrane M, Sullivan KM, Dagnew AF, Curran D, Schuind A. Adjuvanted recombinant zoster vaccine decreases herpes zoster-associated pain and the use of pain medication across 3 randomized, placebo-controlled trials. Pain. 2023 Apr 1;164(4):741-748. doi: 10.1097/j.pain.0000000000002760. Epub 2022 Aug 19. PMID 36066965
- [Derived] Carryn S, Cheuvart B, Povey M, Dagnew AF, Harpaz R, van der Most R, Casabona G. No Consistent Evidence of Decreased Exposure to Varicella-Zoster Virus Among Older Adults in Countries with Universal Varicella Vaccination. J Infect Dis. 2022 Feb 1;225(3):413-421. doi: 10.1093/infdis/jiab500. PMID 34609490
- [Derived] Kim JH, Diaz-Decaro J, Jiang N, Hwang SJ, Choo EJ, Co M, Hastie A, Hui DSC, Irimajiri J, Lee J, Leung EM, Tang H, Tsuru T, Watson P, Wu Z, Yu CJ, Yuan Y, Zahaf T, Cunningham AL, Schuind A. The adjuvanted recombinant zoster vaccine is efficacious and safe in Asian adults >/= 50 years of age: a sub-cohort analysis of the ZOE-50 and ZOE-70 randomized trials. Hum Vaccin Immunother. 2021 Jul 3;17(7):2050-2057. doi: 10.1080/21645515.2020.1859321. Epub 2021 Feb 19. PMID 33606577
- [Derived] Dagnew AF, Rausch D, Herve C, Zahaf T, Levin MJ, Schuind A; ZOE-50/70 study group. Efficacy and serious adverse events profile of the adjuvanted recombinant zoster vaccine in adults with pre-existing potential immune-mediated diseases: a pooled post hoc analysis on two parallel randomized trials. Rheumatology (Oxford). 2021 Mar 2;60(3):1226-1233. doi: 10.1093/rheumatology/keaa424. PMID 32910152
- [Derived] Colindres R, Wascotte V, Brecx A, Clarke C, Herve C, Kim JH, Levin MJ, Oostvogels L, Zahaf T, Schuind A, Cunningham AL. Post hoc analysis of reactogenicity trends between dose 1 and dose 2 of the adjuvanted recombinant zoster vaccine in two parallel randomized trials. Hum Vaccin Immunother. 2020 Nov 1;16(11):2628-2633. doi: 10.1080/21645515.2020.1741312. Epub 2020 Apr 29. PMID 32347767
- [Derived] Willer DO, Oostvogels L, Cunningham AL, Gervais P, Gorfinkel I, Hyung Kim J, Talarico C, Wascotte V, Zahaf T, Colindres R, Schuind A; ZOE 50/70 study groups. Efficacy of the adjuvanted recombinant zoster vaccine (RZV) by sex, geographic region, and geographic ancestry/ethnicity: A post-hoc analysis of the ZOE-50 and ZOE-70 randomized trials. Vaccine. 2019 Oct 8;37(43):6262-6267. doi: 10.1016/j.vaccine.2019.09.028. Epub 2019 Sep 16. PMID 31537443
- [Derived] Lopez-Fauqued M, Campora L, Delannois F, El Idrissi M, Oostvogels L, De Looze FJ, Diez-Domingo J, Heineman TC, Lal H, McElhaney JE, McNeil SA, Yeo W, Tavares-Da-Silva F; ZOE-50/70 Study Group. Safety profile of the adjuvanted recombinant zoster vaccine: Pooled analysis of two large randomised phase 3 trials. Vaccine. 2019 Apr 24;37(18):2482-2493. doi: 10.1016/j.vaccine.2019.03.043. Epub 2019 Mar 29. PMID 30935742
- [Derived] Curran D, Oostvogels L, Heineman T, Matthews S, McElhaney J, McNeil S, Diez-Domingo J, Lal H, Andrews C, Athan E, Berglund J, Campora L, de Looze F, Korhonen T, Leung E, Levin M, Volpi A, Johnson RW; ZOE-50/70 Study Group. Quality of Life Impact of an Adjuvanted Recombinant Zoster Vaccine in Adults Aged 50 Years and Older. J Gerontol A Biol Sci Med Sci. 2019 Jul 12;74(8):1231-1238. doi: 10.1093/gerona/gly150. PMID 29955836
- See also: IPD for this study will be made available via the Clinical Study Data Request site. — https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of all the subjects enrolled into this study, only 15405 received vaccination and were hence considered to start the study.
Groups:
- GSK1437173A Group: Subjects received herpes zoster subunit vaccine (gE/AS01B vaccine: GSK1437173A) according to a 0, 2-month schedule.
- Placebo Group: Subjects received saline solution (NaCl solution) as control according to a 0, 2-month schedule.
Period: Overall Study
Arm/Group | GSK1437173A Group | Placebo Group
Started | 7695 | 7710
Completed | 6773 | 6808
Not Completed | 922 | 902
Not completed — Serious Adverse Event | 227 | 235
Not completed — Withdrawal by Subject | 368 | 354
Not completed — Protocol Violation | 19 | 21
Not completed — Non-serious adverse event | 30 | 18
Not completed — Other unspecified reasons | 47 | 35
Not completed — Suspected HZ episode | 0 | 2
Not completed — Lost to Follow-up | 183 | 194
Not completed — Migrated/ moved from study area | 48 | 43

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK1437173A Group | Placebo Group | Total
Number analyzed (Participants) | 7695 | 7710 | 15405
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.4 (9.0) | 62.3 (9.0) | 62.35 (9.0)
Age, Customized [Count of Participants; unit: Participants]
  50 - 59 YOA | 3644 | 3642 | 7286
  60 - 69 YOA | 2243 | 2245 | 4488
  >= 70 YOA | 1808 | 1823 | 3631
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4709 | 4711 | 9420
  Male | 2986 | 2999 | 5985

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Confirmed Herpes Zoster (HZ) Cases
Description: Confirmed HZ cases during the study were assessed in the Modified Total Vaccinated Cohort (mTVc)
Time Frame: During the entire study period (3 to 5 year period following Day 0)
Population: The analysis was based on the modified total vaccinated cohort, which included subjects from the total vaccinated cohort, except those who were not administered with the second vaccination or who developed a confirmed case of Herpes Zoster prior to 1 month after the second vaccination.
Measure: Count of Participants; unit: Participants
Groups:
- GSK1437173A 50-59 YOA Group: Subjects aged between 50 and 59 years of age (YOA), receiving the GSK1437173A vaccine according to a 0, 2-month schedule.
- GSK1437173A 60-69 YOA Group: Subjects aged between 60 and 69 years of age (YOA), receiving the GSK1437173A vaccine according to a 0, 2-month schedule.
- GSK1437173A Over 70 YOA Group: Subjects aged above 70 years of age (YOA), receiving the GSK1437173A vaccine according to a 0, 2-month schedule.
- GSK1437173A Overall Ages Group: Subjects aged over 50 years of age (YOA), receiving the GSK1437173A vaccine according to a 0, 2-month schedule.
- Placebo 50-59 YOA Group: Subjects aged between 50 and 59 years of age (YOA), receiving placebo according to a 0, 2-month schedule.
- Placebo 60-69 YOA Group: Subjects aged between 60 and 69 years of age (YOA), receiving placebo according to a 0, 2-month schedule.
- Placebo Over 70 YOA Group: Subjects aged above 70 years of age (YOA), receiving placebo according to a 0, 2-month schedule.
- Placebo Overall Ages Group: Subjects aged over 50 years of age (YOA), receiving placebo according to a 0, 2-month schedule.
Arm/Group | GSK1437173A 50-59 YOA Group | GSK1437173A 60-69 YOA Group | GSK1437173A Over 70 YOA Group | GSK1437173A Overall Ages Group | Placebo 50-59 YOA Group | Placebo 60-69 YOA Group | Placebo Over 70 YOA Group | Placebo Overall Ages Group
Number analyzed (Participants) | 3492 | 2141 | 1711 | 7344 | 3525 | 2166 | 1724 | 7415
Participants | 3 | 2 | 1 | 6 | 87 | 75 | 48 | 210
Statistical Analysis 1: Comparison: GSK1437173A 50-59 YOA Group vs Placebo 50-59 YOA Group; Comparison of vaccine efficacy in prevention of HZ between GSK1437173A 50-59 YOA group and placebo 50-59 YOA group; Test type: Other — Criteria for the vaccine efficacy (VE) objective of herpes zoster subunit (HZ/su) vaccine against herpes zoster (HZ) disease, in the 50-59 YOA strata : The lower limit (LL) of the two-sided 95% confidence interval (CI) of VE had to be above 10%; p < 0.0001, Poisson exact test — Two sided exact P-value conditional to number of cases; Vaccine efficacy = 96.6, 95% CI 2-sided [89.6 to 99.3]
Statistical Analysis 2: Comparison: GSK1437173A 60-69 YOA Group vs Placebo 60-69 YOA Group; Comparison of vaccine efficacy in prevention of HZ between GSK1437173A over 60-69 YOA group and placebo over 60-69 YOA group; Test type: Other — Criteria for the VE objective of HZ/su vaccine against herpes zoster disease, in the 60-69 YOA strata : The lower limit (LL) of the two-sided 95% confidence interval (CI) of VE had to be above 10%; p < 0.0001, Poisson exact test — Two sided exact P-value conditional to number of cases; Vaccine efficacy = 97.4, 95% CI 2-sided [90.1 to 99.7]
Statistical Analysis 3: Comparison: GSK1437173A Over 70 YOA Group vs Placebo Over 70 YOA Group; Comparison of vaccine efficacy in prevention of HZ between GSK1437173A over 70 YOA group and placebo over 70 YOA group; Test type: Other — Criteria for the VE objective of HZ/su vaccine against herpes zoster disease, in the 70-79 YOA strata : The lower limit (LL) of the two-sided 95% confidence interval (CI) of VE had to be above 10%; p = 0.0001, Poisson exact test — Two sided exact P-value conditional to number of cases; Vaccine efficacy = 97.9, 95% CI 2-sided [87.9 to 100]
Statistical Analysis 4: Comparison: GSK1437173A Overall Ages Group vs Placebo Overall Ages Group; Comparison of vaccine efficacy in prevention of HZ between GSK1437173A overall ages group and placebo overall ages group; Test type: Other — Criteria for the VE objective of HZ/su vaccine against herpes zoster disease, in the overall age strata : The lower limit (LL) of the two-sided 95% confidence interval (CI) of VE had to be above 10%; p < 0.0001, Poisson exact test — Two sided exact P-value conditional to number of cases; Vaccine efficacy = 97.2, 95% CI 2-sided [93.7 to 99]

2. Secondary Outcome: Number of Subjects With Any Episodes of Post-Herpetic Neuralgia (PHN)
Description: The incidence of PHN was calculated using the modified total vaccinated chort.
Time Frame: During the entire study period (3 to 5 year period following Day 0)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A 50-59 YOA Group | GSK1437173A 60-69 YOA Group | GSK1437173A Over 70 YOA Group | GSK1437173A Overall Ages Group | Placebo 50-59 YOA Group | Placebo 60-69 YOA Group | Placebo Over 70 YOA Group | Placebo Overall Ages Group
Number analyzed (Participants) | 3491 | 2140 | 1709 | 7430 | 3523 | 2166 | 1724 | 7413
Participants | 0 | 0 | 0 | 0 | 8 | 2 | 8 | 18
Statistical Analysis 1: Comparison: GSK1437173A 50-59 YOA Group vs Placebo 50-59 YOA Group; Comparison of vaccine efficacy in prevention of PHN between GSK1437173A 50-59 YOA group and placebo 50-59 YOA group; Test type: Other — Criteria for the VE objective of HZ/su vaccine against PHN in the 50-59 YOA strata: The lower limit of the 95% CI of VE had to be above 0%; p = 0.0081, Poisson exact test; Vaccine efficacy = 100, 95% CI 2-sided [40.9 to 100]
Statistical Analysis 2: Comparison: GSK1437173A 60-69 YOA Group vs Placebo 60-69 YOA Group; Comparison of vaccine efficacy in prevention of PHN between GSK1437173A 60-69 YOA group and placebo 60-69 YOA group; Test type: Other — Criteria for VE objective of HZ/su vaccine against PHN in the 60-69 YOA strata: The lower limit of the 95% CI of VE had to be above 0%; p = 0.5097, Poisson exact test; Vaccine efficacy = 100, 95% CI 2-sided [-442.8 to 100]
Statistical Analysis 3: Comparison: GSK1437173A Over 70 YOA Group vs Placebo Over 70 YOA Group; Comparison of vaccine efficacy in prevention of PHN between GSK1437173A over 70 YOA group and placebo over 70 YOA group; Test type: Other — Criteria for the VE objective of HZ/su vaccine against PHN in the 70-79 YOA strata: The lower limit of the 95% CI of VE had to be above 0%; p = 0.0078, Poisson exact test; Vaccine efficacy = 100, 95% CI 2-sided [41.4 to 100]
Statistical Analysis 4: Comparison: GSK1437173A Overall Ages Group vs Placebo Overall Ages Group; Comparison of vaccine efficacy in prevention of PHN between GSK1437173A overall ages group and placebo overall ages group; Test type: Other — Criteria for the VE objective of HZ/su vaccine against PHN in the overall ages strata: The lower limit of the 95% CI of VE had to be above 0%; p < 0.0001, Poisson exact test; Vaccine efficacy = 100, 95% CI 2-sided [77.1 to 100]

3. Secondary Outcome: Number of Subjects With a Reduction of Duration of Severe 'Worst' HZ-associated Pain
Description: Severe 'worst' pain was defined as HZ-associated pain rated as 3 or above on the 'worst pain' Zoster Brief Pain Inventory (ZBPI) questionnaire. The outcome assessed the duration of severe 'worst' HZ-associated pain following the onset of a confirmed HZ rash over the entire pain reporting period as measured by the ZBPI in subjects with confirmed HZ. This analysis involved any subject reporting clinically significant pain (i.e. pain with a score of 3 or more on a 0-10 point scale) at any time during the study.
Time Frame: During the entire study period (3 to 5 year period following Day 0)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A 50-59 YOA Group | GSK1437173A 60-69 YOA Group | GSK1437173A Over 70 YOA Group | GSK1437173A Overall Ages Group | Placebo 50-59 YOA Group | Placebo 60-69 YOA Group | Placebo Over 70 YOA Group | Placebo Overall Ages Group
Number analyzed (Participants) | 4 | 3 | 2 | 9 | 103 | 90 | 61 | 254
Participants | 4 | 1 | 2 | 7 | 91 | 74 | 56 | 221

4. Secondary Outcome: Number of Subjects With Confirmed HZ Episode Related Mortality
Description: The analysis focused on the number of subjects who died due to HZ
Time Frame: During the entire study period (3 to 5 year period following Day 0)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A 50-59 YOA Group | GSK1437173A 60-69 YOA Group | GSK1437173A Over 70 YOA Group | GSK1437173A Overall Ages Group | Placebo 50-59 YOA Group | Placebo 60-69 YOA Group | Placebo Over 70 YOA Group | Placebo Overall Ages Group
Number analyzed (Participants) | 3491 | 2140 | 1709 | 7340 | 3523 | 2166 | 1724 | 7413
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Subjects With HZ Related Complications
Description: The analysis focused on the incidence of HZ complications in subjects with confirmed HZ
Time Frame: During the entire study period (3 to 5 year period following Day 0)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A 50-59 YOA Group | GSK1437173A 60-69 YOA Group | GSK1437173A Over 70 YOA Group | GSK1437173A Overall Ages Group | Placebo 50-59 YOA Group | Placebo 60-69 YOA Group | Placebo Over 70 YOA Group | Placebo Overall Ages Group
Number analyzed (Participants) | 4 | 3 | 2 | 9 | 103 | 90 | 61 | 254
Participants | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 6

6. Secondary Outcome: Number of Subjects With Confirmed HZ Episode Related Hospitalizations
Description: The analysis focused on confirmed HZ episode related hospitalizations.
Time Frame: During the entire study period (3 to 5 year period following Day 0)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A 50-59 YOA Group | GSK1437173A 60-69 YOA Group | GSK1437173A Over 70 YOA Group | GSK1437173A Overall Ages Group | Placebo 50-59 YOA Group | Placebo 60-69 YOA Group | Placebo Over 70 YOA Group | Placebo Overall Ages Group
Number analyzed (Participants) | 3491 | 2140 | 1709 | 7340 | 3523 | 2166 | 1724 | 7413
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Subjects With a Confirmed HZ Episode Having a Reduction of Duration of Pain Medication Associated With HZ
Description: The analysis focused on patients who experienced a reduction in duration of pain medication administered for HZ in subjects with confirmed HZ.
Time Frame: During the entire study period (3 to 5 year period following Day 0)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A 50-59 YOA Group | GSK1437173A 60-69 YOA Group | GSK1437173A Over 70 YOA Group | GSK1437173A Overall Ages Group | Placebo 50-59 YOA Group | Placebo 60-69 YOA Group | Placebo Over 70 YOA Group | Placebo Overall Ages Group
Number analyzed (Participants) | 4 | 3 | 2 | 9 | 103 | 90 | 61 | 254
Participants | 3 | 2 | 1 | 6 | 82 | 63 | 45 | 190

8. Secondary Outcome: Number of Subjects With a Confirmed HZ Episode Taking Pain Medication Associated With HZ
Description: The analysis focused on subjects taking pain medication due to HZ
Time Frame: During the entire study period (3 to 5 year period following Day 0)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A 50-59 YOA Group | GSK1437173A 60-69 YOA Group | GSK1437173A Over 70 YOA Group | GSK1437173A Overall Ages Group | Placebo 50-59 YOA Group | Placebo 60-69 YOA Group | Placebo Over 70 YOA Group | Placebo Overall Ages Group
Number analyzed (Participants) | 4 | 3 | 2 | 9 | 103 | 90 | 61 | 254
Participants | 3 | 2 | 1 | 6 | 82 | 63 | 45 | 190

9. Secondary Outcome: Number of Days With Severe 'Worst' HZ-associated Pain.
Description: Severe 'worst' pain was defined as HZ-associated pain rated as 3 or above on the 'worst pain' ZBPI questionnaire. This Outcome Measure was only assessed participants with confirmed HZ. This analysis involved any subject reporting ZBPI clinically significant pain (i.e. pain with a score of 3 or more on a 0-10 point scale) at any time during the study.
Time Frame: During the entire study period (3 to 5 year period following Day 0)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | GSK1437173A 50-59 YOA Group | GSK1437173A 60-69 YOA Group | GSK1437173A Over 70 YOA Group | GSK1437173A Overall Ages Group | Placebo 50-59 YOA Group | Placebo 60-69 YOA Group | Placebo Over 70 YOA Group | Placebo Overall Ages Group
Number analyzed (Participants) | 4 | 1 | 2 | 7 | 91 | 74 | 56 | 221
Days | 12.0 (11.8) | 78.0 (0.0) | 9.0 (4.2) | 20.6 (26.8) | 28.7 (48.4) | 21.6 (29.3) | 44.0 (74.4) | 30.2 (51.9)

10. Secondary Outcome: Number of Subjects With Confirmed HZ Episode Related Mortality and Hospitalizations
Description: The analysis focused on confirmed HZ episode related hospitalizations and deaths.
Time Frame: During the entire study period (3 to 5 year period following Day 0)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A 50-59 YOA Group | GSK1437173A 60-69 YOA Group | GSK1437173A Over 70 YOA Group | GSK1437173A Overall Ages Group | Placebo 50-59 YOA Group | Placebo 60-69 YOA Group | Placebo Over 70 YOA Group | Placebo Overall Ages Group
Number analyzed (Participants) | 3491 | 2140 | 1709 | 7340 | 3523 | 2166 | 1724 | 7413
Participants
  Mortality | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hospitalization | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Mortality or hospitalization | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Number of Subjects With HZ Related Complications, by Complication Type
Description: Complication types included HZ vasculitis, Disseminated Disease, Ophtalmic Disease, Neurologic Disease, Visceral Disease and Stroke. This Outcome Measure was only assessed participants with confirmed HZ.
Time Frame: During the entire study period (3 to 5 year period following Day 0)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A 50-59 YOA Group | GSK1437173A 60-69 YOA Group | GSK1437173A Over 70 YOA Group | GSK1437173A Overall Ages Group | Placebo 50-59 YOA Group | Placebo 60-69 YOA Group | Placebo Over 70 YOA Group | Placebo Overall Ages Group
Number analyzed (Participants) | 4 | 3 | 2 | 9 | 103 | 90 | 61 | 254
Participants
  At least one complication | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 6
  HZ vasculitis | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Disseminated Disease | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 4
  Ophtalmic Disease | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Neurologic Disease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Visceral Disease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Stroke | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Distribution of Pain Medication Associated With HZ
Description: The distribution of pain medication included 1 to 3 or more separate medications. This Outcome Measure was only assessed on participants with confirmed HZ.
Time Frame: During the entire study period (3 to 5 year period following Day 0)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A 50-59 YOA Group | GSK1437173A 60-69 YOA Group | GSK1437173A Over 70 YOA Group | GSK1437173A Overall Ages Group | Placebo 50-59 YOA Group | Placebo 60-69 YOA Group | Placebo Over 70 YOA Group | Placebo Overall Ages Group
Number analyzed (Participants) | 4 | 3 | 2 | 9 | 103 | 90 | 61 | 254
Participants
  At least one pain medication | 3 | 2 | 1 | 6 | 82 | 63 | 45 | 190
  1 pain medication only | 1 | 1 | 0 | 2 | 30 | 23 | 14 | 67
  2 pain medications only | 1 | 1 | 0 | 2 | 26 | 19 | 9 | 54
  3 pain medications or more | 1 | 0 | 1 | 2 | 26 | 21 | 22 | 69

13. Secondary Outcome: Number of Days of Pain Medication Associated With HZ
Description: The analysis was performed on subjects with a confirmed HZ episode
Time Frame: During the entire study period (3 to 5 year period following Day 0)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | GSK1437173A 50-59 YOA Group | GSK1437173A 60-69 YOA Group | GSK1437173A Over 70 YOA Group | GSK1437173A Overall Ages Group | Placebo 50-59 YOA Group | Placebo 60-69 YOA Group | Placebo Over 70 YOA Group | Placebo Overall Ages Group
Number analyzed (Participants) | 3 | 2 | 1 | 6 | 82 | 63 | 45 | 190
Days | 17.3 (14.5) | 20.5 (16.3) | 63.0 (0.0) | 26.0 (21.6) | 49.2 (121.5) | 74.3 (166.3) | 127.7 (266.9) | 76.1 (181.5)

14. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = Significant pain at rest that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site. Relationship analysis was not performed.
Time Frame: During the 7-day (Days 0-6) post-vaccination period
Population: The analysis was performed on the total vaccinated cohort - Diary Card, which was a subset of subjects from the total vaccinated cohort, who completed diary cards with any solicited symptoms during the 7 days (Day 0 to Day 6) post vaccination period.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 4379 | 4375
Participants
  Any Pain, Dose 1: number analyzed (Participants) | 4359 | 4361
  Any Pain, Dose 1 | 3120 | 352
  Grade 3 Pain, Dose 1: number analyzed (Participants) | 4359 | 4361
  Grade 3 Pain, Dose 1 | 159 | 6
  Any Redness, Dose 1: number analyzed (Participants) | 4359 | 4361
  Any Redness, Dose 1 | 1225 | 40
  Grade 3 Redness, Dose 1: number analyzed (Participants) | 4359 | 4361
  Grade 3 Redness, Dose 1 | 82 | 0
  Any Swelling, Dose 1: number analyzed (Participants) | 4359 | 4361
  Any Swelling, Dose 1 | 810 | 31
  Grade 3 Swelling, Dose 1: number analyzed (Participants) | 4359 | 4361
  Grade 3 Swelling, Dose 1 | 28 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 4207 | 4224
  Any Pain, Dose 2 | 2807 | 258
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 4207 | 4224
  Grade 3 Pain, Dose 2 | 185 | 10
  Any Redness, Dose 2: number analyzed (Participants) | 4207 | 4224
  Any Redness, Dose 2 | 1151 | 24
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 4207 | 4224
  Grade 3 Redness, Dose 2 | 56 | 0
  Any Swelling, Dose 2: number analyzed (Participants) | 4207 | 4224
  Any Swelling, Dose 2 | 762 | 17
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 4207 | 4224
  Grade 3 Swelling, Dose 2 | 18 | 0
  Any Pain, Overall | 3463 | 490
  Grade 3 Pain, Overall | 293 | 16
  Any Redness, Overall | 1665 | 59
  Grade 3 Redness, Overall | 121 | 0
  Any Swelling, Overall | 1153 | 46
  Grade 3 Swelling, Overall | 43 | 0

15. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, GI (gastrointestinal) symptoms (included nausea, vomiting, diarrhoea and/or abdominal pain), fever [defined as oral, axillary, rectal or tympanic temperature equal to or above 37.5 degrees Celsius (°C)], headache, myalgia, shivering and sweating. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = temperature> 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: Within the 7-day (Days 0-6) post-vaccination period
Population: The analysis was performed on the TVc - Diary Card, which was a subset of subjects from the TVc, who completed diary cards with any solicited symptoms during the 7 days (Day 0 to Day 6) post vaccination period.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 4372 | 4376
Participants
  Any Fatigue, Dose 1: number analyzed (Participants) | 4346 | 4362
  Any Fatigue, Dose 1 | 1395 | 531
  Grade 3 Fatigue, Dose 1: number analyzed (Participants) | 4346 | 4362
  Grade 3 Fatigue, Dose 1 | 109 | 29
  Related fatigue, Dose 1: number analyzed (Participants) | 4346 | 4362
  Related fatigue, Dose 1 | 1153 | 355
  Any GI symptoms, Dose 1: number analyzed (Participants) | 4346 | 4362
  Any GI symptoms, Dose 1 | 465 | 263
  Grade 3 GI symptoms, Dose 1: number analyzed (Participants) | 4346 | 4362
  Grade 3 GI symptoms, Dose 1 | 30 | 12
  Related GI symptoms, Dose 1: number analyzed (Participants) | 4346 | 4362
  Related GI symptoms, Dose 1 | 317 | 141
  Any Headache, Dose 1: number analyzed (Participants) | 4346 | 4362
  Any Headache, Dose 1 | 1112 | 511
  Grade 3 Headache, Dose 1: number analyzed (Participants) | 4346 | 4362
  Grade 3 Headache, Dose 1 | 67 | 20
  Related Headache, Dose 1: number analyzed (Participants) | 4346 | 4362
  Related Headache, Dose 1 | 891 | 341
  Any Myalgia, Dose 1: number analyzed (Participants) | 4346 | 4362
  Any Myalgia, Dose 1 | 1446 | 377
  Grade 3 Myalgia, Dose 1: number analyzed (Participants) | 4346 | 4362
  Grade 3 Myalgia, Dose 1 | 104 | 21
  Related Myalgia, Dose 1: number analyzed (Participants) | 4346 | 4362
  Related Myalgia, Dose 1 | 1231 | 265
  Any Shivering, Dose 1: number analyzed (Participants) | 4346 | 4362
  Any Shivering, Dose 1 | 632 | 166
  Grade 3 Shivering, Dose 1: number analyzed (Participants) | 4346 | 4362
  Grade 3 Shivering, Dose 1 | 69 | 3
  Related Shivering, Dose 1: number analyzed (Participants) | 4346 | 4362
  Related Shivering, Dose 1 | 539 | 104
  Any Temperature, Dose 1: number analyzed (Participants) | 4346 | 4362
  Any Temperature, Dose 1 | 500 | 65
  Grade 3 Temperature, Dose 1: number analyzed (Participants) | 4346 | 4362
  Grade 3 Temperature, Dose 1 | 7 | 1
  Related Temperature, Dose 1: number analyzed (Participants) | 4346 | 4362
  Related Temperature, Dose 1 | 420 | 38
  Any Fatigue, Dose 2: number analyzed (Participants) | 4205 | 4222
  Any Fatigue, Dose 2 | 1456 | 379
  Grade 3 Fatigue, Dose 2: number analyzed (Participants) | 4205 | 4222
  Grade 3 Fatigue, Dose 2 | 157 | 18
  Related fatigue, Dose 2: number analyzed (Participants) | 4205 | 4222
  Related fatigue, Dose 2 | 1270 | 279
  Any GI symptoms, Dose 2: number analyzed (Participants) | 4205 | 4222
  Any GI symptoms, Dose 2 | 495 | 183
  Grade 3 GI symptoms, Dose 2: number analyzed (Participants) | 4205 | 4222
  Grade 3 GI symptoms, Dose 2 | 33 | 14
  Related GI symptoms, Dose 2: number analyzed (Participants) | 4205 | 4222
  Related GI symptoms, Dose 2 | 392 | 91
  Any Headache, Dose 2: number analyzed (Participants) | 4205 | 4222
  Any Headache, Dose 2 | 1249 | 340
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 4205 | 4222
  Grade 3 Headache, Dose 2 | 105 | 13
  Related Headache, Dose 2: number analyzed (Participants) | 4205 | 4222
  Related Headache, Dose 2 | 1107 | 219
  Any Myalgia, Dose 2: number analyzed (Participants) | 4205 | 4222
  Any Myalgia, Dose 2 | 1474 | 274
  Grade 3 Myalgia, Dose 2: number analyzed (Participants) | 4205 | 4222
  Grade 3 Myalgia, Dose 2 | 160 | 13
  Related Myalgia, Dose 2: number analyzed (Participants) | 4205 | 4222
  Related Myalgia, Dose 2 | 1314 | 197
  Any Shivering, Dose 2: number analyzed (Participants) | 4205 | 4222
  Any Shivering, Dose 2 | 947 | 128
  Grade 3 Shivering, Dose 2: number analyzed (Participants) | 4205 | 4222
  Grade 3 Shivering, Dose 2 | 139 | 9
  Related Shivering, Dose 2: number analyzed (Participants) | 4205 | 4222
  Related Shivering, Dose 2 | 838 | 88
  Any Temperature, Dose 2: number analyzed (Participants) | 4205 | 4222
  Any Temperature, Dose 2 | 645 | 72
  Grade 3 Temperature, Dose 2: number analyzed (Participants) | 4205 | 4222
  Grade 3 Temperature, Dose 2 | 8 | 5
  Related Temperature, Dose 2: number analyzed (Participants) | 4205 | 4222
  Related Temperature, Dose 2 | 571 | 40
  Any Fatigue, Overall | 2006 | 728
  Grade 3 Fatigue, Overall | 241 | 46
  Related fatigue, Overall | 1724 | 522
  Any GI symptoms, Overall | 787 | 386
  Grade 3 GI symptoms, Overall | 61 | 25
  Related GI symptoms, Overall | 591 | 206
  Any Headache, Overall | 1714 | 700
  Grade 3 Headache, Overall | 157 | 30
  Related Headache, Overall | 1470 | 469
  Any Myalgia, Overall | 2023 | 529
  Grade 3 Myalgia, Overall | 236 | 31
  Related Myalgia, Overall | 1791 | 390
  Any Shivering, Overall | 1232 | 259
  Grade 3 Shivering, Overall | 192 | 11
  Related Shivering, Overall | 1082 | 177
  Any Temperature, Overall | 940 | 132
  Grade 3 Temperature, Overall | 14 | 6
  Related Temperature, Overall | 813 | 78

16. Secondary Outcome: Number of Subjects With Any and Grade 3 Symptoms (Solicited and Unsolicited)
Description: Number of subjects with any and grade 3 solicited and unsolicited symptoms were tabulated
Time Frame: Within the 7-day (Days 0-6) post-vaccination period
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 4457 | 4464
Participants
  Any solicited or unsolicited symptoms | 3766 | 1691
  Grade 3 solicited or unsolicited symptoms | 759 | 145

17. Secondary Outcome: Number of Subjects With Any and Related Potential Immune Mediated Diseases (pIMDs)
Description: Occurrence and relationship to vaccination of any potential immune-mediated diseases (pIMDs) in all subjects
Time Frame: During the entire study period (3 to 5 year period following Day 0)
Population: This analysis was based on the the total vaccinated cohort, which included all subjects with at least one dose of study vaccine or placebo administered.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 7695 | 7710
Participants
  Any pIMDs | 87 | 105
  Related pIMDs | 8 | 12

18. Secondary Outcome: Number of Subjects With AEs With Any and Related Medically Attended Visit
Description: Occurrence and relationship to vaccination of medically attended visits (defined as hospitalizations, emergency room visits or visits to or from medical personnel), other than routine health care visits in all subjects.
Time Frame: From Month 0 to Month 8 post-vaccination
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 7695 | 7710
Participants
  Any medically attended visits | 2952 | 3072
  Related medically attended visits | 142 | 60

19. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: Occurrence, intensity and relationship to vaccination of unsolicited AEs, according to the Medical Dictionary for Regulatory Activities (MedDRA) classification in all subjects An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: Within 30 days (Days 0 - 29) after each vaccination
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 7695 | 7710
Participants
  Any unsolicited AEs | 3534 | 2426
  Grade 3 unsolicited AEs | 609 | 298
  Related unsolicited AEs | 2199 | 439

20. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Occurrence and relationship to vaccination of all SAEs in all subjects. Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: Within the 30-day (Days 0-29) post-vaccination period, up to Month 14 and up to study end (3 to 5 year period following Day 0)
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 7695 | 7710
Participants
  Any SAEs (up to Day 30) | 88 | 97
  Related SAEs (up to Day 30) | 1 | 3
  Any SAEs (up to Month 14) | 594 | 590
  Related SAEs (up to Month 14) | 3 | 6
  Any SAEs (up to study end) | 727 | 731
  Related SAEs (up to study end) | 3 | 7

21. Secondary Outcome: Number of Subjects With SAEs Related to Study Participation or to a Concurrent GSK Medication/Vaccine
Description: The number of subjects with SAEs related to study participation or to a concurrent GSK medication/vaccine were tabulated
Time Frame: During the entire study period (3 to 5 year period following Day 0)
Population: The analysis was based on TVC, which included all subjects with at least one dose of the study vaccine or place administered.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 7695 | 7710
Participants | 43 | 25

22. Secondary Outcome: Number of Subjects With Fatal SAEs
Description: Number of subjects with fatal SAEs during the entire study period were tabulated
Time Frame: During the entire study period (3 to 5 years following day 0)
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 7695 | 7710
Participants | 208 | 221

ADVERSE EVENTS:
Time Frame: Solicited symptoms: within 7 days post-vaccination Unsolicited AEs: within 30 days post vaccination SAEs: during the entire study period (3 to 5 year period following Day 0)
Arm/Group | GSK1437173A Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 11/7695 | 15/7710
Serious Adverse Events (participants affected / at risk) | 727/7695 | 731/7710
Other Adverse Events (participants affected / at risk) | 5586/7695 | 1893/7710
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK1437173A Group (N=7695) | Placebo Group (N=7710)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 4 (4)
Anaemia vitamin b12 deficiency (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (3) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Splenic haemorrhage (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 4 (4) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 8 (8) | 19 (19)
Angina pectoris (Cardiac disorders) | 3 (4) | 3 (3)
Angina unstable (Cardiac disorders) | 2 (2) | 4 (4)
Aortic valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 2 (2)
Arrhythmia (Cardiac disorders) | 6 (6) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 19 (23) | 6 (6)
Atrial flutter (Cardiac disorders) | 4 (4) | 4 (4)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 1 (1) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 2 (2)
Atrioventricular block second degree (Cardiac disorders) | 2 (2) | 0 (0)
Bradyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 2 (2) | 2 (2)
Cardiac arrest (Cardiac disorders) | 8 (8) | 8 (8)
Cardiac failure (Cardiac disorders) | 20 (21) | 24 (27)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 3 (3)
Cardiac failure chronic (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 14 (15) | 10 (10)
Cardiac valve disease (Cardiac disorders) | 2 (2) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 2 (2)
Cardiogenic shock (Cardiac disorders) | 3 (3) | 1 (1)
Cardiomyopathy alcoholic (Cardiac disorders) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 1 (1)
Cardiovascular deconditioning (Cardiac disorders) | 0 (0) | 1 (1)
Cardiovascular insufficiency (Cardiac disorders) | 1 (1) | 0 (0)
Cor pulmonale (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 11 (11) | 17 (19)
Coronary artery insufficiency (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 4 (4) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 2 (2) | 0 (0)
Left ventricular failure (Cardiac disorders) | 3 (3) | 0 (0)
Mitral valve prolapse (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 28 (28) | 27 (27)
Myocardial ischaemia (Cardiac disorders) | 7 (7) | 11 (11)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 2 (2) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 2 (2) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 3 (3) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cystic fibrosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Hernia congenital (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Hypertrophic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Odontogenic cyst (Cardiac disorders) | 0 (0) | 1 (1)
Deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Motion sickness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 4 (4) | 3 (3)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Basedow's disease (Endocrine disorders) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 1 (1) | 0 (0)
Hypopituitarism (Endocrine disorders) | 1 (1) | 0 (0)
Thyroiditis subacute (Endocrine disorders) | 1 (1) | 0 (0)
Amaurosis fugax (Eye disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 2 (2) | 5 (5)
Eyelid ptosis (Eye disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Lens dislocation (Eye disorders) | 0 (0) | 1 (1)
Macular cyst (Eye disorders) | 0 (0) | 1 (1)
Macular hole (Eye disorders) | 0 (0) | 1 (1)
Neovascular age-related macular degeneration (Eye disorders) | 0 (0) | 1 (1)
Retinal artery occlusion (Eye disorders) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1) | 4 (4)
Retinal tear (Eye disorders) | 0 (0) | 1 (1)
Vitreous detachment (Eye disorders) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal strangulated hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 3 (3) | 1 (1)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Enterovesical fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric mucosal lesion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 3 (3) | 3 (3)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastritis (Gastrointestinal disorders) | 5 (5) | 4 (4)
Gastritis alcoholic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3) | 4 (4)
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gingival disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 4 (4)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 3 (3)
Ileus (Gastrointestinal disorders) | 1 (1) | 3 (3)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 3 (3) | 8 (8)
Intestinal congestion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 3 (3) | 3 (3)
Intestinal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 2 (2)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 4 (4)
Mallory-weiss syndrome (Gastrointestinal disorders) | 1 (1) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pancreatic cyst (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatic fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 4 (4) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 5 (5) | 6 (7)
Pancreatitis necrotising (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peptic ulcer perforation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peritoneal cyst (Gastrointestinal disorders) | 1 (1) | 1 (1)
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumoperitoneum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Portal hypertensive gastropathy (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 3 (3)
Splenic artery aneurysm (Gastrointestinal disorders) | 0 (0) | 1 (1)
Subileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Volvulus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 3 (3) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 12 (12) | 10 (12)
Death (General disorders) | 11 (11) | 15 (15)
Device dislocation (General disorders) | 0 (0) | 1 (1)
Device failure (General disorders) | 0 (0) | 1 (1)
Drowning (General disorders) | 1 (1) | 1 (1)
Drug withdrawal syndrome (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 1 (1)
Gravitational oedema (General disorders) | 1 (1) | 0 (0)
Hernia (General disorders) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 2 (2) | 0 (0)
Multi-organ failure (General disorders) | 6 (6) | 2 (2)
Non-cardiac chest pain (General disorders) | 2 (2) | 1 (1)
Pain (General disorders) | 1 (1) | 2 (2)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
Polyp (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 1 (1)
Strangulated hernia (General disorders) | 0 (0) | 1 (1)
Sudden cardiac death (General disorders) | 0 (0) | 3 (3)
Sudden death (General disorders) | 5 (5) | 7 (7)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 3 (3)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 5 (5) | 6 (6)
Cholecystitis acute (Hepatobiliary disorders) | 6 (6) | 4 (4)
Cholelithiasis (Hepatobiliary disorders) | 7 (7) | 10 (10)
Fatty liver alcoholic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Gallbladder polyp (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary dyskinesia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 2 (2) | 1 (1)
Sarcoidosis (Immune system disorders) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Abdominal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Abscess neck (Infections and infestations) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1)
Appendiceal abscess (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 3 (3) | 6 (6)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 2 (2)
Bacteriuria (Infections and infestations) | 1 (1) | 0 (0)
Biliary sepsis (Infections and infestations) | 0 (0) | 1 (1)
Breast abscess (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 3 (3) | 4 (4)
Bronchitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Bronchopneumonia (Infections and infestations) | 2 (2) | 0 (0)
Candiduria (Infections and infestations) | 0 (0) | 1 (1)
Catheter site infection (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 8 (8) | 6 (6)
Cellulitis orbital (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Chronic sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 2 (2) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 3 (3)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Cystitis klebsiella (Infections and infestations) | 0 (0) | 1 (1)
Dengue fever (Infections and infestations) | 0 (0) | 1 (1)
Diabetic gangrene (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 4 (4) | 6 (7)
Encephalomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1) | 1 (1)
Endometritis (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 2 (2) | 3 (3)
Fungaemia (Infections and infestations) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 3 (3) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (4) | 4 (4)
Gastroenteritis caliciviral (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis clostridial (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis salmonella (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Helicobacter gastritis (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis a (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Infected dermal cyst (Infections and infestations) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 1 (1)
Infectious colitis (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 1 (1) | 0 (0)
Labyrinthitis (Infections and infestations) | 1 (1) | 0 (0)
Leptospirosis (Infections and infestations) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0)
Lobar pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 6 (6)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Lymph node tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Meningitis pneumococcal (Infections and infestations) | 0 (0) | 1 (1)
Mycobacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Nasal abscess (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Neuroborreliosis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 4 (5) | 2 (2)
Osteomyelitis chronic (Infections and infestations) | 0 (0) | 1 (1)
Otitis media chronic (Infections and infestations) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 2 (2)
Peritonsillar abscess (Infections and infestations) | 1 (1) | 0 (0)
Pertussis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 40 (41) | 26 (28)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia mycoplasmal (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 0 (0) | 3 (3)
Pseudomembranous colitis (Infections and infestations) | 2 (2) | 1 (1)
Pyelonephritis (Infections and infestations) | 6 (6) | 3 (3)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 2 (2)
Respiratory tract infection (Infections and infestations) | 3 (3) | 2 (2)
Sepsis (Infections and infestations) | 7 (7) | 13 (14)
Septic shock (Infections and infestations) | 1 (1) | 4 (4)
Serratia infection (Infections and infestations) | 1 (1) | 0 (0)
Shigella infection (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis fungal (Infections and infestations) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 2 (2) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1)
Subdiaphragmatic abscess (Infections and infestations) | 0 (0) | 1 (1)
Superinfection (Infections and infestations) | 1 (1) | 0 (0)
Testicular abscess (Infections and infestations) | 1 (1) | 0 (0)
Toxic shock syndrome (Infections and infestations) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1)
Tularaemia (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2)
Upper respiratory tract infection bacterial (Infections and infestations) | 2 (2) | 0 (0)
Urethritis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 10 (10) | 10 (10)
Urosepsis (Infections and infestations) | 2 (2) | 3 (3)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 1 (1)
Viral sepsis (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Visceral leishmaniasis (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 2 (2) | 0 (0)
Wound infection pseudomonas (Infections and infestations) | 1 (1) | 1 (1)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Aneurysm perforation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 7 (7) | 4 (4)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Burns third degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cataract operation complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Chemical poisoning (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Comminuted fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Concussion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Electrical burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Eye penetration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Femoral neck fracture (Injury, poisoning and procedural complications) | 5 (5) | 4 (5)
Femur fracture (Injury, poisoning and procedural complications) | 7 (7) | 3 (3)
Fibula fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Flail chest (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fractured sacrum (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Gun shot wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Head injury (Injury, poisoning and procedural complications) | 3 (3) | 4 (4)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 6 (6)
Humerus fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Incarcerated incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Nerve root injury cervical (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Open fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Pubis fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 7 (7) | 7 (7)
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 5 (5)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Snake bite (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Spinal cord injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Splenic rupture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Sternal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 3 (4) | 1 (1)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Traumatic shock (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Vascular pseudoaneurysm ruptured (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anticoagulation drug level above therapeutic (Investigations) | 0 (0) | 1 (1)
Blood heavy metal increased (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperammonaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 4 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 7 (7)
Joint destruction (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 8 (8) | 11 (11)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Soft tissue mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Still's disease adult onset (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Acute promyelocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adult t-cell lymphoma/leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Angioimmunoblastic t-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1)
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign neoplasm of orbit (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign soft tissue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bile duct adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 5 (5)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (4)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 6 (6)
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Bronchial neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carcinoid tumour of the small bowel (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Cervix carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 11 (11)
Diffuse large b-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Extranodal marginal zone b-cell lymphoma (malt type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Fallopian tube cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 4 (4)
Gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Glomus tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 4 (4)
Invasive papillary breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Laryngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 3 (3)
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Lung adenocarcinoma stage i (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (11) | 6 (6)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Malignant neoplasm of pleura metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Metastases to lymph (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Metastases to pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0)
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Ovarian fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 8 (9)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Phaeochromocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Pleural mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 9 (9)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Renal oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small intestine adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Spinal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Testicular neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Amyotrophic lateral sclerosis (Nervous system disorders) | 2 (2) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Basal ganglia haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Basal ganglia infarction (Nervous system disorders) | 1 (1) | 0 (0)
Brain injury (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery disease (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 1 (1)
Carotid artery thrombosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 2 (2) | 4 (4)
Cerebral infarction (Nervous system disorders) | 8 (8) | 6 (7)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 19 (19) | 12 (12)
Cerebrovascular disorder (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular insufficiency (Nervous system disorders) | 1 (1) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Chronic inflammatory demyelinating polyradiculoneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Coma (Nervous system disorders) | 0 (0) | 1 (1)
Dementia alzheimer's type (Nervous system disorders) | 0 (0) | 1 (1)
Demyelinating polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 1 (2) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 4 (4)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1) | 4 (4)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 0 (0)
Guillain-barre syndrome (Nervous system disorders) | 1 (1) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhagic transformation stroke (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 3 (3)
Ivth nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Lacunar infarction (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 2 (2)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Mononeuritis (Nervous system disorders) | 0 (0) | 1 (1)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 1 (1)
Myelopathy (Nervous system disorders) | 0 (0) | 1 (1)
Nerve compression (Nervous system disorders) | 1 (1) | 0 (0)
Nervous system disorder (Nervous system disorders) | 1 (1) | 0 (0)
Neuritis cranial (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Paraneoplastic neurological syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Post polio syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 1 (1)
Radiculopathy (Nervous system disorders) | 0 (0) | 2 (2)
Reversible ischaemic neurological deficit (Nervous system disorders) | 1 (1) | 0 (0)
Ruptured cerebral aneurysm (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 2 (2) | 1 (1)
Seizure (Nervous system disorders) | 3 (3) | 3 (3)
Spinal claudication (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 2 (2) | 4 (4)
Syncope (Nervous system disorders) | 8 (8) | 8 (8)
Transient global amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 8 (8) | 6 (7)
Trigeminal neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Vascular encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Vasculitis cerebral (Nervous system disorders) | 1 (1) | 0 (0)
Viith nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Abnormal behaviour (Psychiatric disorders) | 0 (0) | 1 (1)
Adjustment disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 4 (4) | 4 (4)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Delirium febrile (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 3 (3) | 4 (4)
Generalised anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Korsakoff's syndrome (Psychiatric disorders) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 3 (3)
Somatoform disorder (Psychiatric disorders) | 2 (2) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 4 (4) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 8 (8) | 4 (4)
Azotaemia (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder prolapse (Renal and urinary disorders) | 0 (0) | 1 (1)
Calculus bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Calculus ureteric (Renal and urinary disorders) | 4 (4) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 2 (2) | 6 (6)
Diabetic nephropathy (Renal and urinary disorders) | 2 (2) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 2 (2)
Renal artery arteriosclerosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal artery occlusion (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal cyst (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal failure (Renal and urinary disorders) | 0 (0) | 3 (3)
Renal impairment (Renal and urinary disorders) | 1 (1) | 1 (1)
Stress urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 2 (2) | 0 (0)
Urethral polyp (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 4 (4)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 3 (3) | 2 (2)
Cystocele (Reproductive system and breast disorders) | 3 (3) | 0 (0)
Endometrial hypertrophy (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Fibrocystic breast disease (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Rectocele (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine enlargement (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterovaginal prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 5 (7)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 8 (10)
Dyspnoea (Reproductive system and breast disorders) | 3 (3) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pickwickian syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural calcification (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary bulla (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 13 (13)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 12 (12)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Leukoplakia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Cardiac pacemaker replacement (Surgical and medical procedures) | 0 (0) | 1 (1)
Aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Angiodysplasia (Vascular disorders) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 3 (3)
Aortic dilatation (Vascular disorders) | 0 (0) | 1 (1)
Aortic dissection (Vascular disorders) | 1 (1) | 0 (0)
Aortic rupture (Vascular disorders) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 0 (0) | 3 (3)
Arterial disorder (Vascular disorders) | 1 (1) | 0 (0)
Arterial thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 1 (1) | 2 (2)
Bleeding varicose vein (Vascular disorders) | 1 (1) | 0 (0)
Circulatory collapse (Vascular disorders) | 2 (2) | 3 (3)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 5 (5)
Diabetic vascular disorder (Vascular disorders) | 1 (2) | 0 (0)
Essential hypertension (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 3 (3)
Haemodynamic instability (Vascular disorders) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 8 (8) | 10 (11)
Hypertensive crisis (Vascular disorders) | 2 (2) | 3 (3)
Hypertensive emergency (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 2 (2)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 3 (3)
Intermittent claudication (Vascular disorders) | 0 (0) | 2 (2)
Orthostatic hypertension (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 2 (2) | 2 (3)
Peripheral arterial occlusive disease (Vascular disorders) | 2 (2) | 4 (4)
Peripheral artery stenosis (Vascular disorders) | 2 (2) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Peripheral embolism (Vascular disorders) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 1 (1)
Peripheral venous disease (Vascular disorders) | 2 (2) | 0 (0)
Polyarteritis nodosa (Vascular disorders) | 0 (0) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 1 (1)
Temporal arteritis (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 2 (2) | 0 (0)
Varicose ulceration (Vascular disorders) | 1 (1) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK1437173A Group (N=7695) | Placebo Group (N=7710)
Gastrointestinal disorder (Gastrointestinal disorders) | 792 (967) | 389 (449)
Chills (General disorders) | 1464 (1860) | 276 (314)
Fatigue (General disorders) | 2211 (3111) | 770 (961)
Injection site erythema (General disorders) | 493 (636) | 10 (11)
Injection site pain (General disorders) | 1390 (2090) | 104 (118)
Injection site swelling (General disorders) | 401 (515) | 6 (6)
Pain (General disorders) | 3575 (6064) | 505 (627)
Pyrexia (General disorders) | 1498 (1839) | 168 (176)
Swelling (General disorders) | 1154 (1573) | 46 (48)
Myalgia (Musculoskeletal and connective tissue disorders) | 2277 (3234) | 571 (704)
Headache (Nervous system disorders) | 2167 (3044) | 929 (1198)
Erythema (Skin and subcutaneous tissue disorders) | 1690 (2408) | 69 (75)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.